CLINICAL TRIAL: NCT06788730
Title: The Effect of Transtheoretical Model Based Healthy Internet Use Programme Supported by Mindfulness Exercise on Problematic Internet Use, Social Skills and Self-Efficacy Levels of Adolescents
Brief Title: The Effect of Transtheoretical Model Based Healthy Internet Use Programme on Problematic Internet Use, Social Skills and Self-Efficacy Level
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B-DEMİRDAĞ
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-05

CONDITIONS: Problematic Internet Use; Behaviour Change
Keywords: Adolescent; Problematic internet use; Mindfulness; Transtheoretical model; Self-efficacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Healthy Internet Use Programme will be carried out as one session per week for 8 weeks. The training programme will be carried out by dividing the students into 2 groups (the first group is 18 and the second group is 19 people). The training programme will be applied to the groups two days in the same week at the times determined by the guidance teacher. Interventions will be applied to the intervention group with trainings, homework applications and interventions to increase healthy internet use.
  Interventions: Behavioral: Transtheoretical Model Based Healthy Internet Use Programme Intervention Supported by Mindfulness Exercise Applied to Adolescents
- Control Group (No Intervention): There will be no intervention. The 37 students in the intervention groups will be followed up for 8 weeks and will not receive any training. The final test will be administered at the end of the eighth week

INTERVENTIONS:
Behavioral: Transtheoretical Model Based Healthy Internet Use Programme Intervention Supported by Mindfulness Exercise Applied to Adolescents — Transtheoretical Model Based Healthy Internet Use Programme Supported by Mindfulness Exercise will be carried out as one session per week for 8 weeks. The training programme will be carried out by dividing the students into 2 groups (the first group is 18 and the second group is 19 people). The training programme will be applied to the groups two days in the same week at the times determined by the guidance teacher. Interventions will be applied to the intervention group with trainings, homework applications and interventions to increase healthy internet use.
  Arms: Intervention Group

SUMMARY:
Adolescence is an important developmental stage to promote positive behaviours and prevent psychological difficulties. Internet addiction problems are more common among children and adolescents worldwide. During adolescence, when many changes such as maturation and gaining autonomy are experienced, the internet is used to escape from responsibilities in life and to cope with adaptation problems. Internet addiction brings many different problems such as changing behavioural changes, deterioration in social functions, and decrease in academic success. For this reason, psychosocial and model-based interventions are important in reducing adolescents' internet addiction and ensuring safe internet use. It is emphasised that behavioural interventions and awareness practices should be started at an early age to reduce problematic internet use (Ding & Li,.2023). Since adolescents spend most of their time at school, schools are very important for the acquisition of healthy behaviours (Throuvala, et al. 2019; Yeun & Han, 2016). Providing access to students in schools is necessary to reach more students and prepare a suitable learning environment (Throuvala, et al 2019). When the literature is examined, it is proven that school-based programmes are effective for adolescents to develop positive behaviours on various issues (Spaas et al 2023; Grande et al 2023). Especially in schools, it is necessary to support healthy internet use and self-efficacy with awareness studies that will prevent adolescents' internet addiction through educational programmes. TTM or mindfulness programmes applied to different age groups have been found to be effective in reducing internet use problems (Chang et al 2023; Hafez et al 2023). However, school-based studies on reducing problematic internet use in Turkey are very few. It is important to conduct school-based internet addiction studies in order to benefit science and society in terms of this deficiency in Turkey. In this study, it was aimed to determine the effect of Transtheoretical (Behaviour Change) Model and Mindfulness-Based Healthy Internet Use Programme on problematic internet use, social skills and self-efficacy levels of adolescents. This study aims to determine the effect of Transtheoretical Model Based Healthy Internet Use Programme Supported by Mindfulness Exercise on Problematic Internet Use, Social Skills and Self-Efficacy Level. This research is a randomised controlled study designed in experimental type, pre-test post-test design. The research will be conducted in Namık Kemal Secondary School in Meram district of Konya province. The sample group was determined as 37 intervention and 37 control groups, totalling 66 students. The pre-test data of the intervention and control groups will be collected by the researcher in the classroom environment before the programme starts and the post-test data will be collected after the programme is completed. In order to determine the sociodemographic characteristics of the students and to form appropriate groups, the Personal Information Form created by the researcher will be used to determine the Internet addiction levels of the students, the Internet Addiction Scale will be used to determine the Internet addiction levels of the students, the Self-Efficacy Scale for Children and the Social Emotional Learning Skills Scale will be used to evaluate the self-efficacy of the students. In the study, data will be collected in two stages (pre-test and post-test) based on self-report with a face-to-face questionnaire form in the classroom environment. At the end of the programme, it is expected that students' internet addiction will decrease and their social support and self-efficacy levels will increase.

ELIGIBILITY:
Inclusion Criteria:

* To be between 13-15 years old
* Knowing Turkish
* Those who scored 50 points or more on the internet addiction scale
* Volunteering to participate in the research
* Parental consent

Exclusion Criteria:

* Participants in a similar accompanying programme

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Problematic Internet Use Scale Score | 1-3 months
  Using the Problematic Internet Use Scale (PIUQ), changes in problematic internet use levels before and after the intervention will be evaluated. The change aims to measure the effect of mindfulness exercises and transtheoretical model based programme in the intervention group.
Change in Self-Efficacy Scale Score | 1-3 months
  Self-efficacy levels will be measured with the General Self-Efficacy Scale (GSES) and the effects of the programme on adolescents' self-efficacy perception will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Kto Karatay University, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want you to share